CLINICAL TRIAL: NCT06783933
Title: Artificial Intelligence-assisted Diagnosis of Congenital Heart Diseases on Chest X-ray
Brief Title: Artificial Intelligence-assisted Diagnosis
Acronym: AID
Status: Active, not recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Beijing Anzhen Hospital (Other); Nanjing Medical University (Other); Shanghai Jiao Tong University School of Medicine (Other); Capital Medical University (Other); Sichuan University (Other); Kunming Medical University (Other); Anhui Medical University (Other); Shandong University (Other); Zhejiang University (Other); Peking Union Medical College (Other); Harbin Medical University (Other); Xi'an Jiaotong University (Other); Huazhong University of Science and Technology (Other); Guangdong Provincial People's Hospital (Other); Wuhan University (Other); Central South University (Other); University of Chinese Academy of Sciences (Unknown); The First Hospital of Hebei Medical University (Other); Handan First Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Anyang Maternal and Child Health Care Center (Unknown); Wenzhou Medical University (Other); Guangxi Medical University (Other); Xinjiang Medical University (Other); Chongqing General Hospital (Other); Tibet Autonomous Region People's Hospital (Other); The Affiliated Hospital of Zunyi Medical College (Unknown); Second Affiliated Hospital of Nanchang University (Other); Second Xiangya Hospital of Central South University (Other); Second Hospital of Shanxi Medical University (Other); Handan Central Hospital (Other); Affiliated First Hospital of Ningxia Medical University (Unknown); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Xijing Hospital (Other); Inner Mongolia People's Hospital (Other); Qinghai province cardiovascular and cerebrovascular disease specialist hospital (Unknown); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); China Medical University, China (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Qilu Hospital of Shandong University (Other); Tianjin Medical University General Hospital (Other); Hainan General Hospital (Other); Fujian Medical University (Other); Lanzhou University Second Hospital (Other); Second Hospital of Jilin University (Other); Zunyi Medical College (Other); Ningxia Medical University (Other); LanZhou University (Other); Jilin University (Other); West China Hospital (Other); Peking University (Other); Fudan University (Other); Ruijin Hospital (Other); Zhengzhou University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-4; 2021YFF0501400 (Other: Ministry of Science and Technology)
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-01

CONDITIONS: Congenital Heart Disease (CHD); Structural Heart Disease
Keywords: artificial intelligence；congenital heart diseases；Chest X-ray；diagnosis
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Previous data of chest X-ray in patients with CHD: Phase 1: Previous data of chest X-ray in patients with CHD. A minimum of 5000 patients is reached.
  Interventions: Diagnostic Test: surgical or interventional validation
- Prospective inclusion of general patients with chest X-ray: Prospective inclusion of general patients with chest X-ray. A minimum of 50000 patients is reached.
  Interventions: Diagnostic Test: surgical or interventional validation

INTERVENTIONS:
Diagnostic Test: surgical or interventional validation — surgical or interventional validation

SUMMARY:
This study aims to investigate whether an AI-assisted decision support can improve the diagnosis of congenital heart diseases on Chest X-ray.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is a structural abnormality of the heart and/or great vessels and the frequency of CHD is nearly 1% in general population. In clinical practice, Chest X-ray is an important routine method for detection of CHD. However, its learning curve is high. Based on Chest X-ray, Artificial intelligence (AI) has the potential to improve the efficiency and accuracy of CHD. This study aims to investigate whether an AI-assisted decision support can improve the diagnosis of congenital heart diseases on Chest X-ray.

This study will enroll subjects with CHD, and the enrollment will be divided into two phases.

Phase 1: Previous data of chest X-ray in patients with CHD. A minimum of 5000 patients is reached.

Phase 2: Prospective inclusion of general patients with chest X-ray. A minimum of 50000 patients is reached.

ELIGIBILITY:
Inclusion Criteria:

1. Chest X-ray of patients with ASD;
2. Chest X-ray of patients with VSD;
3. Chest X-ray of patients with PDA;
4. Chest X-ray of patients with PFO;
5. Chest X-ray of patients with PS;
6. Chest X-ray of patients with TOF/PAA;
7. Chest X-ray of patients with MS;
8. Chest X-ray of patients with other heart diseases;

Exclusion Criteria:

1. CHD Patients without surgical, interventional validation;
2. Serious Scoliosis;
3. Pulmonary inflammation or consolidation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll subjects with CHD and structural heart diseases.
Sampling Method: Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2030-01-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
accuracy with AI-assisted diagnosis | 12 months
  Number of subjects with accuracy of CHD ; based on surgical validation or interventional validation.

CONTACTS AND LOCATIONS:
Overall Officials: Shihua Zhao, MD and PhD, Study Chair — Fuwai Hospital, Beijing, China
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author upon reasonable request.